CLINICAL TRIAL: NCT04151823
Title: Effect of POSTbiotics Supplementation on Microbiome in OBese Children: the POST-OB Study
Acronym: POST-OB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Elvira Verduci, Principal Investigator, Paediatrician, University of Milan Researcher, University of Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/ST/135-2
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Childhood Obesity
Keywords: Childhood obesity; Nutrition; Gut microbiota; Postbiotics
MeSH Terms: conditions — Pediatric Obesity | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postbiotic &vitamin D3, lifestyle intervention. (Experimental): Postbiotics will be given at the dose of 80 mg/day (2 ml per day SMART D3 MATRIX Smartfarma S.r.l. Via San Vittore 40 - 20123 MILAN; immunofos from Lactobacillus paracasei CNCM I-5220). 2 mL of product will give 1600 UI/die of VIT D3. Healthy living habits will be encouraged at t0, t1 and t2 visit.
  Interventions: Drug: Vitamin D3; Drug: Immunofos; Other: Promotion of physical activity; Other: Healthy food habits promotion

INTERVENTIONS:
Drug: Vitamin D3 — 2 ml per day SMART D3 MATRIX Smartfarma S.r.l. Via San Vittore 40 - 20123 MILAN: 2 mL of product will give 1600 UI/die of VIT D3.
Drug: Immunofos — Postbiotics will be given at the dose of 80 mg/day. immunofos from Lactobacillus paracasei CNCM I-5220).
Other: Promotion of physical activity — Promotion of physical activity will be encouraged at t0, t1, t2
Other: Healthy food habits promotion — Promotion of healthy food habits will be encouraged at t0, t1, t2

SUMMARY:
This study evaluates the possible effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, on gut microbiota composition and metabolite production. It also wants to determine whether postbiotics supplementation, combined with interventions to improve diet and lifestyle, reduces adverse metabolic consequences together with their co-morbidities.

All participants will follow a behaviour (promotion of physical activity) and dietary treatment according to Italian dietary guidelines for childhood obesity.

Postbiotics and vitamin D3 will be given orally for four months; patients will be evaluated four months after supplementation and diet-lifestyle intervention and four months after the end of supplementation and after the alone diet-lifestyle intervention with blood testing and echosonography of the liver.

DETAILED DESCRIPTION:
25-30 Caucasian obese children will be enrolled at the Pediatric Department of San Paolo Hospital - University of Milan.

Stool samples from all enrolled patients at the different time points (t0, before supplementation and diet-lifestyle intervention, t1, four months after supplementation and diet-lifestyle intervention and t2 four months after the end of supplementation and after the alone diet-lifestyle intervention) will be collected and stored at -80°C until the following investigation:

1. study of the microbiota biodiversity by high-throughput sequencing techniques (16S rRNA gene sequencing) in order to establish whether postbiotics could modulate the microbial composition in obese children;
2. analysis of short chain fatty acids concentration by gas-chromatography (GC-FID) in order to monitor the effect of postbiotics intake modulating microbial metabolite production.

The following tasks will be also performed at t0, t1 and t2:

* Clinical examination including: physical examination, Tanner score evaluation; Bristol Stool Chart
* Blood pressure will be checked in all children by using oscillometric devices validated in the pediatric age group.
* Anthropometry including body circumferences and skinfolds, calculation of BMI z scores and body composition. Body composition will be assessed using an air displacement plethysmography system (BOD POD COSMED-USA).
* Dietary assessment:

  1. Food intakes will be recorded by prospective 3-d weighed food records obtained with food scales. Parents will be advised on how to record all food and beverages consumed during 2 weekdays and 1 weekend day. Quantification and analysis of the energy intake and nutrient composition will be performed with an ad hoc PC software (MètaDieta®, Me.Te.Da S.r.l., San Benedetto del Tronto, Italy).
  2. Mediterranean Diet Quality Index (KIDMED) questionnaire for Mediterranean Diet assessment. The KIDMED index ranges from 0 to 12, and is based on a 16-question test that can be self-administered. The sums of the values from the administered test will be classified into three levels:

     1. 8 or more: optimal Mediterranean diet;
     2. 4-7: improvement needed to adjust intake to Mediterranean patterns.
     3. 3 or less: very low diet quality.
* Hematological and biochemical status including:

  1. Complete cell blood count;
  2. Metabolic and nutritional parameters according to local routines for childhood obesity (fasting glucose, fasting insulin, LDL, HDL, total cholesterol, triglycerides, Apolipoprotein A and Apolipoprotein B levels, transaminases and amma-glutamyl transferase). Oral Glucose Tolerance Test (OGTT) will be performed. The insulin sensitivity and insulin resistance was assessed by calculating HOMA index (Homeostasis Model Assessment) and QUICKI (Quantitative Insulin-Sensitivity Check Index), using the following formulas:

     * HOMA: fasting plasma insulin in mU/l x FPG in mmol/l/22.5
     * QUICKI: 1/(log10 fasting plasma insulin in mU/l + log10 glucose in mg/dl)
  3. Inflammatory index (VES, high-sensitive CRP, including fecal calprotectin)
* Liver ultrasonography will be performed by a single evaluator.

All participants will follow a behavior (promotion of physical activity) and dietary treatment according to Italian dietary guidelines for childhood obesity.

Postbiotics will be given at the dose of 80 mg/day (2 ml per day SMART D3 MATRIX Smartfarma S.r.l. Via San Vittore 40 - 20123 MILAN; fermented fructooligosaccharides from Lactobacillus paracasei strain CNCM I-5220). 2 mk of product will give 1600 UI/die of VIT D3.

ELIGIBILITY:
Inclusion Criteria:

* 6 <Age <14 years
* Severe obesity (>3 DS) according to WHO classification.
* Gestational age: 37-42 weeks.
* Birth-weight: > 2500 g e < 4000 g
* Caucasian

Exclusion Criteria:

* secondary obesity
* supplementation with pre/probiotics (in the previous 3 months);
* antibiotic treatment (in the previous 3 months);
* chronic or acute intestinal diseases (in the previous 3 months).

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-01-07 (Estimated); Study Completion 2021-01-07 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiota composition | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in short chain fatty acids production by gut microbiota | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).

SECONDARY OUTCOMES:
Changes in HDL-cholesterol levels | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in LDL-cholesterol levels | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in triglycerides levels | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in systemic arterial blood pressure | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in body mass index | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in Bristol stool chart | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in puberal stage | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in fasting glucose levels | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in fasting insulin levels | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in oral glucose tolerance test results | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in Apoprotein A1 levels | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in Apoprotein B levels | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in alanine aminotransferase (ALT) levels | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in aspartate aminotransferase (AST) levels | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in Gamma-glutamyl transferase (GGT) levels | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in complete cell blood count | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in total cholesterol levels | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in Homeostasis Model Assessment (HOMA) index | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in Quantitative Insulin-Sensitivity Check Index (QUICKI) | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in erythrocyte sedimentation rate (ESR) | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in C-reactive protein (CRP) levels | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in fecal calprotectin levels | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Echosonographic changes in liver morphology (degree of steatosis) | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in body mass composition assessed with air displacement plethysmography system | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in body circumference (waist, left arm) | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).
Changes in body skinfold thickness (waist, posterior skinfold and anterior skinfold of left arm) | t0: 0 t1: +4 months t2: +8 months
  Effect of postbiotics supplementation, combined with interventions aimed at improving diet and lifestyle, will be evaluated. Difference in gut microbiota composition will be evaluated before starting supplementation (t0), at the end of supplementation (t1: +4 months) e after 4 months of dietary dietary-lifestyle intervention without supplementation (t2: +8 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Paolo, Milan, Italy

IPD SHARING:
Plan to Share IPD: No